CLINICAL TRIAL: NCT01611272
Title: A Post Marketing Surveillance to Evaluate the Safety and Efficacy of Brilinta
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5130L00019
Record Dates: First submitted 2012-05-25; First posted 2012-06-04 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Acute Coronary Syndromes
Keywords: Unstable angina
MeSH Terms: conditions — Acute Coronary Syndrome; Angina, Unstable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Unstable angina, Non ST-segment Elevation Myocardial Infarction or ST-segment elevation myocardial infarction including patients managed medically, and those who are managed with percutaneous coronary intervention or coronary artery by-pass grafting

SUMMARY:
To identify the following items through the post marketing surveillance under routine clinical practice after marketing authorization of Brilinta Tablet: the occurrence of unrevealed Serious Adverse Events (SAEs), current status of occurrence of Adverse Events (AEs), the factors that may influence safety and efficacy of the drug.

DETAILED DESCRIPTION:
A Post Marketing Surveillance to evaluate the safety and efficacy of Brilinta

ELIGIBILITY:
Inclusion Criteria:

* Patients with Acute Coronary Syndromes
* Patients who are taking ticagrelor and ASA daily(75-150mg), or Patients who are taking ticagrelor only(In the case that the patients have contraindication with ASA. Contraindication should be recorded in accordance with local PI on CRFs)
* Patients who have signed the Data release consent form prior to enrollment in this surveillance

Exclusion Criteria:

* Patients with hypersensitivity to ingredients of this drug or with moderate or severe hepatic impairment or with medical history of intracranial hemorrhage
* Patients with pathological hemorrhage at the time of administration
* Patients being administrated strong CYP3A4 inhibitors

Ages: 19 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who take Brilinta according to the local approval condition
Sampling Method: Probability Sample
Enrollment: 3402 (Actual)
Dates: Start 2013-04-30 (Actual); Primary Completion 2016-07-20 (Actual); Study Completion 2016-07-20 (Actual)

PRIMARY OUTCOMES:
Number of Hemorrhage events | up to 54 months
Number of other AEs | up to 54 months

SECONDARY OUTCOMES:
Number of Stroke events | up to 54 months
  for efficacy
Number of Cardiovascular (CV) related deaths events | up to 54 months
  for efficacy
Number of Myocardial Infarction events | up to 54 months
  for efficacy

CONTACTS AND LOCATIONS:
Overall Officials: JooWon Lee, Study Director — AstraZeneca Korea
Locations (23):
- South Korea (23):
  - Research Site, Cheonan-si, Chungcheongnam-do
  - Research Site, Chuncheon, Gangwon-do
  - Research Site, Wŏnju, Gangwon-do
  - Research Site, Ansan-si, Gyeonggi-do
  - Research Site, Anyang-si, Gyeonggi-do
  - Research Site, Bucheon-si, Gyeonggi-do
  - Research Site, Goyang-si, Gyeonggi-do
  - Research Site, Koyang-shi, Gyeonggi-do
  - Research Site, Seongnam-si, Gyeonggi-do
  - Research Site, Suwon, Gyeonggi-do
  - Research Site, Andong, Gyeongsangbuk-do
  - Research Site, Gumi, Gyeongsangbuk-do
  - Research Site, Gimhae, Gyeongsangnam-do
  - Research Site, Iksan-si, Jeollabuk-do
  - Research Site, Jeonju, Jeollabuk-do
  - Research Site, Suncheon-si, Jeollanam-do
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Gwangju
  - Research Site, Incheon
  - Research Site, Seoul
  - Research Site, Ulsan

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=487&filename=CSR_Synopsis.pdf